CLINICAL TRIAL: NCT00780247
Title: Environmental Influences on Vitamin D Status
Acronym: Alaska/Hawaii
Status: Completed | Type: Observational
Sponsor: Creighton University (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Laura Armas, M D, Creighton University
Other Study IDs: Creighton6; WIRB approval 20080712
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Last update posted 2008-10-27 (Estimated); Status verified 2008-10

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D; Sun; Latitude; Vitamin D status
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Alaska residents: 50 "healthy" community dwelling males or females.
- Hawaiian residents: 50 "healthy" community dwelling males or females at each site

SUMMARY:
Vitamin D deficiency is a common problem. The principal source of vitamin D for humans is solar exposure, with cutaneous synthesis of vitamin D by photoconversion of 7-dehydrocholesterol in the skin to pre-vitamin D3. Latitude, altitude, season, skin pigmentation, and age are recognized factors that influence how much vitamin D can be made by solar exposure. However, the relative influences of each are largely unknown and we cannot reliably answer the question of how much sun exposure an individual needs at various latitudes and at various seasons in order to ensure normal vitamin D status.

DETAILED DESCRIPTION:
Purpose of the study: To determine the effect of environmental influences on Vitamin D status.

Specific Aims

1. To measure the prevailing 25D and Vitamin D levels in communities at diverse latitudes (Alaska and Hawaii).
2. To collect information on variables that influence Vitamin D status such as skin color, history of sun exposure and sunscreen use, diet history, vitamin and calcium supplements used, and BMI.
3. To collect typical food samples from the region for future analysis of their Vitamin D and 25D content.
4. To collect a blood sample for DNA analysis of inter-individual differences in Vitamin D metabolism (Gc or Vitamin D binding protein alleles).

ELIGIBILITY:
Inclusion Criteria:

* Able to consent and come for a study visit. Male or female males and females ages 18-60.

Exclusion Criteria:

* Unable to consent or come to a visit, taking Vitamin D supplements, anticonvulsants, barbiturates, steroids, having granulomatous disease, or liver or kidney disease as these medications and conditions interfere with Vitamin D metabolism.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Age of Subjects: The subjects will be between ages 18-60. The upper age is limited to age 60 as aging skin is less able to make vitamin D, therefore a separate study of elderly people would be more appropriate.
  Racial and Ethnic Origin: Both sites have a diverse ethnic and racial population and the subjects will be as representative of the population as possible.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To measure the prevailing 25D and Vitamin D levels in communities at diverse latitudes | crosssectional

SECONDARY OUTCOMES:
2. To collect information on variables that influence Vitamin D status such to collect information on skin color, history of sun exposure and sunscreen use, diet history, vitamin and calcium supplements used, and BMI. | cross sectional
To collect a blood sample for DNA analysis of inter-individual differences in Vitamin D metabolism (Gc or Vitamin D binding protein alleles). | cross sectional

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Armas, MD, Principal Investigator — Creighton University
Locations (1):
- Alaska Kidney and Diabetes Associates, Anchorage, Alaska, United States